CLINICAL TRIAL: NCT02506062
Title: A Randomized, Single-blinded Placebo-controlled Trial of Ischemic Preconditioning in Raynaud's Phenomenon (RP)
Brief Title: A Trial of Ischemic Preconditioning in Raynaud's Phenomenon (RP)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Janet Pope, Principal Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 106798
Record Dates: First submitted 2015-07-08; First posted 2015-07-22 (Estimated); Last update posted 2018-08-08 (Actual); Status verified 2018-08

CONDITIONS: Raynaud Disease; Raynaud's Phenomenon
Keywords: ischemic preconditioning; Raynaud's Phenomenon; (RP)
MeSH Terms: conditions — Raynaud Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active Arm - 200 mmHg (Experimental): Patients who start in the active arm of the study will receive ischemic preconditioning (IPC) treatment consisting of applying the blood pressure cuff to a pressure of 200 mmHg for 2 minutes and thirty seconds with a resting period of two minutes and thirty seconds between treatments. This procedure is performed four times, for a total of twenty minutes per treatment. This treatment will be done three times a week. Patients may choose to treat at home with a portable manual blood pressure machine or may be treated in clinic by research staff. Patients will receive treatment for two weeks followed by a wash-out period (no treatment) of two weeks. Patients will then receive the placebo treatment. This completes their participation in the study.
  Interventions: Device: Manual blood pressure cuff inflation over brachial artery
- Placebo Arm - 60 mmHg (Placebo Comparator): Patients who start in the placebo arm will receive placebo treatment, consisting of applying the blood pressure cuff to a pressure of 60 mmHg for 2 minutes and thirty seconds with a resting period of two minutes and thirty seconds between treatments. This procedure is performed four times, for a total of twenty minutes per treatment. This treatment will be done three times a week for two weeks followed by a two week wash-out and then two weeks in the active treatment phase, thus completing their participation in the study.
  Interventions: Device: Manual blood pressure cuff inflation over brachial artery

INTERVENTIONS:
Device: Manual blood pressure cuff inflation over brachial artery — A manual blood pressure cuff (sphygmomanometer) is used in the study as a tourniquet in order to perform a controlled, consistent level of ischemia (200mmHg/active arm or 60 mmHg/placebo arm).

SUMMARY:
This trial will test the efficacy of brief periods of controlled limb ischemia (remote ischemic preconditioning, RIPC) as an effective treatment of patients with Raynaud's Phenomenon (RP).The hypothesis of this trial is that due to its vasoprotective effects, RIPC would be more effective than placebo in the treatment of both primary and secondary RP, as defined by decreased frequency, duration, and severity of attacks. This trial was also designed to monitor the tolerance of RIPC in a rheumatologic population. Patients will not be required to stop any current treatment for RP.

DETAILED DESCRIPTION:
Raynaud's phenomenon (RP) is defined as vasospasms of arteries causing pallor and at least one other color change upon reperfusion such as cyanosis or redness. The current treatments for RP (channel blockers, PDE5 inhibitors, etc.) have only modest efficacy and are associated with many side-effects including headaches, flushing, hypotension and fluid retention that require stopping the medication. Thus, identification of an innovative treatment is an important therapeutic goal in RP patients.

Ischemic preconditioning is a simple non-invasive procedure which consists of 4 consecutive episodes of brief ischemia caused by placing a pneumatic cuff at the level of the brachial artery and inflating it to 200 mm Hg for 2.5 minutes, followed by 2.5 minutes of reperfusion. Over 20 years IPC has generated tremendous scientific interest being described as the most powerful available form of in vivo protection against ischemic injury.

This clinical trial will measure the efficiency of RIPC in decreasing the frequency, duration and severity of RP attacks. 24 patients will be recruited from the Rheumatology clinic of St. Joseph's Health Care in London, Ontario. As they enter the trial, subjects will be assigned to a treatment or a placebo group according to a pre-set randomization schedule. The trial will be single-blinded (patient).

The primary outcome measures (frequency, duration and severity) will be assessed by the patient on a daily basis using a journal provided by the investigator. Secondary outcome measures will include functions questionnaires (Raynaud's Condition Score, s-HAQ-DI, DASH) and biological markers of endothelial damage (P-selectin, I-CAM, VEGF), will be conducted every two weeks: at baseline, post-placebo, post-washout, and post-treatment phases.

Patients participation will span 8 weeks. The first two weeks are a baseline measurement for the status of RP using the journals, questionnaires, and serum tests. The treatment period will last 6 weeks in which the subject will be completing the arm of the IPC regimen to which he/she has been assigned.

Other results which may arise from the trial are:

* The tolerance of RIPC in rheumatology patients, by monitoring side-effects.
* The attitude of rheumatology patients in using non-pharmacological treatments, by a questionnaire.
* Elucidating parts of the RP mechanism, by measuring bio-markers
* Differences between primary and secondary RP, by stratified randomization

The results will be analyzed for all three primary outcome measures as a difference of between baseline and treatment. These differences will be compared between treatment and placebo and each will be stratified for primary vs. secondary and possibly other demographic data.

This trial, if positive, will offer another treatment to RP patients. This option will possibly have fewer side-effects and be better accepted because it is a common and safe non-pharmacological intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Primary or secondary RP, as diagnosed by a rheumatologist
2. Clinical need for treatment for RP
3. At least 7 RP attacks per week
4. Systolic blood pressure above 80mmHg
5. Willing to provide informed consent

Exclusion Criteria:

1. New or changed dose of drugs used for RP treatment in the last 2 weeks: calcium channel blockers, alpha1-adrenergic blockers, angiotensin II receptor antagonists, nitroglycerin, prostaglandins, pentoxifylline, endothelin antagonists and/or phosphodiesterase type 5 inhibitors.
2. Non-compliance with past therapies

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2015-07; Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Changes in frequency of RP attacks | Entire study duration (8 weeks including pretreatment and washout period)
  The subject will self-assess the number of RP attacks daily in their RP diary.
Changes in severity of RP attacks | Entire study duration (8 weeks including pretreatment and washout period)
  Severity will be evaluated on a scale of 1 to 10. The subject will self-assess the severity in their RP diary. (0 = no difficulty with RP condition, 10 = extreme difficulty with RP condition).
Changes in duration of RP attacks | Entire study duration (8 weeks including pretreatment and washout period)
  The subject will self-assess the duration (in minutes) of RP attacks daily in their RP diary.

SECONDARY OUTCOMES:
Functions questionnaires (Raynaud's Condition Score) | Every 2 weeks at clinic visits (baseline, after intervention, after washout, and after placebo) for a total of 6 weeks
Biological marker of endothelial damage (P-selectin) | Every 2 weeks at clinic visits (baseline, after intervention, after washout, and after placebo) for a total of 6 weeks
Biological marker of endothelial damage (I-CAM) | Every 2 weeks at clinic visits (baseline, after intervention, after washout, and after placebo) for a total of 6 weeks
Biological marker of endothelial damage (VEGF) | Every 2 weeks at clinic visits (baseline, after intervention, after washout, and after placebo) for a total of 6 weeks
Functions questionnaires (HAQ-DI) | Every 2 weeks at clinic visits (baseline, after intervention, after washout, and after placebo) for a total of 6 weeks
  Health Assessment Questionnaire - Disability Index
Functions questionnaires (DASH) | Every 2 weeks at clinic visits (baseline, after intervention, after washout, and after placebo) for a total of 6 weeks
  Disabilities of the Arm, Shoulder, and Hand

CONTACTS AND LOCATIONS:
Overall Officials: Janet E Pope, Principal Investigator — Division of Rheumatology, Department of Medicine, Western University
Locations (1):
- Rheumatology Clinic, St. Joseph's Health Care, London, Ontario, Canada

REFERENCES:
- [Background] Pope J. Raynaud's phenomenon (primary). BMJ Clin Evid. 2013 Oct 10;2013:1119. PMID 24112969
- [Background] Pope JE. The diagnosis and treatment of Raynaud's phenomenon: a practical approach. Drugs. 2007;67(4):517-25. doi: 10.2165/00003495-200767040-00003. PMID 17352512
- [Background] Khan F. Vascular abnormalities in Raynaud's phenomenon. Scott Med J. 1999 Feb;44(1):4-6. doi: 10.1177/003693309904400102. No abstract available. PMID 10218222
- [Background] Thompson AE, Pope JE. Calcium channel blockers for primary Raynaud's phenomenon: a meta-analysis. Rheumatology (Oxford). 2005 Feb;44(2):145-50. doi: 10.1093/rheumatology/keh390. Epub 2004 Nov 16. PMID 15546967
- [Background] Lazaris AM, Maheras AN, Vasdekis SN, Karkaletsis KG, Charalambopoulos A, Kakisis JD, Martikos G, Patapis P, Giamarellos-Bourboulis EJ, Karatzas GM, Liakakos TD. Protective effect of remote ischemic preconditioning in renal ischemia/reperfusion injury, in a model of thoracoabdominal aorta approach. J Surg Res. 2009 Jun 15;154(2):267-73. doi: 10.1016/j.jss.2008.06.037. Epub 2008 Jul 26. PMID 19376531
- [Background] Jensen HA, Loukogeorgakis S, Yannopoulos F, Rimpilainen E, Petzold A, Tuominen H, Lepola P, Macallister RJ, Deanfield JE, Makela T, Alestalo K, Kiviluoma K, Anttila V, Tsang V, Juvonen T. Remote ischemic preconditioning protects the brain against injury after hypothermic circulatory arrest. Circulation. 2011 Feb 22;123(7):714-21. doi: 10.1161/CIRCULATIONAHA.110.986497. Epub 2011 Feb 7. PMID 21300953
- [Background] Tapuria N, Kumar Y, Habib MM, Abu Amara M, Seifalian AM, Davidson BR. Remote ischemic preconditioning: a novel protective method from ischemia reperfusion injury--a review. J Surg Res. 2008 Dec;150(2):304-30. doi: 10.1016/j.jss.2007.12.747. Epub 2008 Jan 22. PMID 19040966
- [Background] Jan WC, Chen CH, Tsai PS, Huang CJ. Limb ischemic preconditioning mitigates lung injury induced by haemorrhagic shock/resuscitation in rats. Resuscitation. 2011 Jun;82(6):760-6. doi: 10.1016/j.resuscitation.2011.02.010. Epub 2011 Mar 12. PMID 21398019
- [Background] Li L, Luo W, Huang L, Zhang W, Gao Y, Jiang H, Zhang C, Long L, Chen S. Remote perconditioning reduces myocardial injury in adult valve replacement: a randomized controlled trial. J Surg Res. 2010 Nov;164(1):e21-6. doi: 10.1016/j.jss.2010.06.016. Epub 2010 Jul 2. PMID 20850778
- [Background] Richard V, Kaeffer N, Tron C, Thuillez C. Ischemic preconditioning protects against coronary endothelial dysfunction induced by ischemia and reperfusion. Circulation. 1994 Mar;89(3):1254-61. doi: 10.1161/01.cir.89.3.1254. PMID 8124814
- [Background] Kharbanda RK, Peters M, Walton B, Kattenhorn M, Mullen M, Klein N, Vallance P, Deanfield J, MacAllister R. Ischemic preconditioning prevents endothelial injury and systemic neutrophil activation during ischemia-reperfusion in humans in vivo. Circulation. 2001 Mar 27;103(12):1624-30. doi: 10.1161/01.cir.103.12.1624. PMID 11273988
- [Background] Davis JM, Gute DC, Jones S, Krsmanovic A, Korthuis RJ. Ischemic preconditioning prevents postischemic P-selectin expression in the rat small intestine. Am J Physiol. 1999 Dec;277(6):H2476-81. doi: 10.1152/ajpheart.1999.277.6.H2476. PMID 10600871
- [Background] Beauchamp P, Richard V, Tamion F, Lallemand F, Lebreton JP, Vaudry H, Daveau M, Thuillez C. Protective effects of preconditioning in cultured rat endothelial cells: effects on neutrophil adhesion and expression of ICAM-1 after anoxia and reoxygenation. Circulation. 1999 Aug 3;100(5):541-6. doi: 10.1161/01.cir.100.5.541. PMID 10430769
- [Background] Jones H, Hopkins N, Bailey TG, Green DJ, Cable NT, Thijssen DH. Seven-day remote ischemic preconditioning improves local and systemic endothelial function and microcirculation in healthy humans. Am J Hypertens. 2014 Jul;27(7):918-25. doi: 10.1093/ajh/hpu004. Epub 2014 Mar 13. PMID 24627443
- [Background] Kimura M, Ueda K, Goto C, Jitsuiki D, Nishioka K, Umemura T, Noma K, Yoshizumi M, Chayama K, Higashi Y. Repetition of ischemic preconditioning augments endothelium-dependent vasodilation in humans: role of endothelium-derived nitric oxide and endothelial progenitor cells. Arterioscler Thromb Vasc Biol. 2007 Jun;27(6):1403-10. doi: 10.1161/ATVBAHA.107.143578. Epub 2007 Apr 19. PMID 17446439
- [Background] Vasdekis SN, Athanasiadis D, Lazaris A, Martikos G, Katsanos AH, Tsivgoulis G, Machairas A, Liakakos T. The role of remote ischemic preconditioning in the treatment of atherosclerotic diseases. Brain Behav. 2013 Nov;3(6):606-16. doi: 10.1002/brb3.161. Epub 2013 Aug 30. PMID 24363964
- [Background] Alreja G, Bugano D, Lotfi A. Effect of remote ischemic preconditioning on myocardial and renal injury: meta-analysis of randomized controlled trials. J Invasive Cardiol. 2012 Feb;24(2):42-8. PMID 22294530
- [Background] Pilcher JM, Young P, Weatherall M, Rahman I, Bonser RS, Beasley RW. A systematic review and meta-analysis of the cardioprotective effects of remote ischaemic preconditioning in open cardiac surgery. J R Soc Med. 2012 Oct;105(10):436-45. doi: 10.1258/jrsm.2012.120049. PMID 23104947
- [Background] Brevoord D, Kranke P, Kuijpers M, Weber N, Hollmann M, Preckel B. Remote ischemic conditioning to protect against ischemia-reperfusion injury: a systematic review and meta-analysis. PLoS One. 2012;7(7):e42179. doi: 10.1371/journal.pone.0042179. Epub 2012 Jul 31. PMID 22860077
- [Background] Li C, Li YS, Xu M, Wen SH, Yao X, Wu Y, Huang CY, Huang WQ, Liu KX. Limb remote ischemic preconditioning for intestinal and pulmonary protection during elective open infrarenal abdominal aortic aneurysm repair: a randomized controlled trial. Anesthesiology. 2013 Apr;118(4):842-52. doi: 10.1097/ALN.0b013e3182850da5. PMID 23353795
- [Background] Koch S, Katsnelson M, Dong C, Perez-Pinzon M. Remote ischemic limb preconditioning after subarachnoid hemorrhage: a phase Ib study of safety and feasibility. Stroke. 2011 May;42(5):1387-91. doi: 10.1161/STROKEAHA.110.605840. Epub 2011 Mar 17. PMID 21415404
- [Background] Luca MC, Liuni A, McLaughlin K, Gori T, Parker JD. Daily ischemic preconditioning provides sustained protection from ischemia-reperfusion induced endothelial dysfunction: a human study. J Am Heart Assoc. 2013 Feb 22;2(1):e000075. doi: 10.1161/JAHA.112.000075. PMID 23525419
- See also: American website of institute of arthritis: general medical information on Raynaud's Disease — http://www.niams.nih.gov/Health_Info/Raynauds_Phenomenon/default.asp